CLINICAL TRIAL: NCT03283501
Title: A Multicenter Observational Registry on Coronary Revascularization After Implantation of Transcatheter Aortic Valve Bioprosthesis
Brief Title: Revascularization After Transcatheter Aortic Valve Implantation (REVIVAL)
Acronym: REVIVAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Enrico Cerrato, Principal Investigator, San Luigi Gonzaga Hospital
Other Study IDs: 001-2017
Record Dates: First submitted 2017-09-04; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Transcatheter Valve Implantation; TAVI
Keywords: TAVI; PCI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PCI after TAVI — Any patient undergoing PCI after TAVI, irrespective of clinical indications and irrespective of whether planned or not at the time of TAVI

SUMMARY:
Evaluate incidence, clinical indications, and feasibility of PCI performed after TAVI.

DETAILED DESCRIPTION:
The increasing operator experience combined with an improved performance of devices have led to extend current transcatheter aortic valve implantation (TAVI) indications to patients at low or intermediate risk. The safety of TAVI in this population was initially tested in small observational studies and recently reported in the randomized PARTNER 2 and Surgical Replacement and Transcatheter Aortic Valve Implantation Trial (SURTAVI) trials, which demonstrated non- inferiority of TAVI in low or intermediate risk patients as compared to surgery with respect to the primary endpoint of death or disabling stroke. In view of the changes in the TAVI population, including younger patients with longer survival, the number of patients that may require coronary revascularization after TAVI is expected to increase over the time. Of note, challenges in performing percutaneous coronary interventions (PCI) in patients previously treated with TAVI have been reported in small series.

Against this background, the purpose of this retrospective multicenter study is to evaluate incidence, clinical indications, and feasibility of PCI performed after TAVI.

Objectives

1. Evaluate the incidence of PCI after TAVI
2. Evaluate the clinical indications for PCI after TAVI
3. Evaluate the technical feasibility of PCI in patients with prior TAVI
4. Evaluate in-hospital and long-term clinical outcomes in patients undergoing PCI after TAVI

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing PCI after TAVI, irrespective of clinical indications and irrespective of whether planned or not at the time of TAVI

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient undergoing PCI after TAVI, irrespective of clinical indications and irrespective of whether planned or not at the time of TAVI
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the incidence of PCI after TAVI | up to 5 year after TAVI implantation
  Evaluate the incidence of PCI after TAVI
Evaluate the clinical indications for PCI after TAVI | intraoperative
  Clinical indication for PCI: stable angina; documented silent ischemia; acute coronary syndrome/non-ST elevation myocardial infarction; acute coronary syndrome/ST elevation myocardial infarction
Evaluate the technical feasibility of PCI in patients with prior TAVI | intraoperative
  Successful target coronary vessel revascularization
Evaluate in-hospital and long-term clinical outcomes in patients undergoing PCI after TAVI | up to 5 year after TAVI implantation
  outcome defined as MACE (Major Adverse Coronary Event) a composite of Death, Myocardial Infarction, Target Lesion Failure

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (2):
  - Humanitas Research Hospital, Humanitas University, Rozzano, Milan
  - Interventional Unit, San Luigi Gonzaga University Hospital, Orbassano, and Rivoli Hospital, Turin, Italy, Turin
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stefanini GG, Cerrato E, Pivato CA, Joner M, Testa L, Rheude T, Pilgrim T, Pavani M, Brouwer J, Lopez Otero D, Munoz Garcia E, Barbanti M, Biasco L, Varbella F, Reimers B, Jimenez Diaz VA, Leoncini M, Salido Tahoces ML, Ielasi A, de la Torre Hernandez JM, Mylotte D, Garot P, Chieffo A, Nombela-Franco L; REVIVAL Investigators. Unplanned Percutaneous Coronary Revascularization After TAVR: A Multicenter International Registry. JACC Cardiovasc Interv. 2021 Jan 25;14(2):198-207. doi: 10.1016/j.jcin.2020.10.031. PMID 33478637
- See also: Organization research website — http://cardiogroup.org